CLINICAL TRIAL: NCT02459509
Title: A Comparison of Two Doses of Intranasal Dexmedetomidine for Premedication in Children - a Double- Blind Randomised Controlled Trial
Brief Title: A Comparison of Two Doses of Intranasal Dexmedetomidine for Premedication in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 15-105
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety, Separation
Keywords: Sedation; dexmedetomidine; pediatric; preoperative period
MeSH Terms: conditions — Anxiety, Separation | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dexmedetomidine 2 mcg/kg (Active Comparator): 2 mcg/kg dexmedetomidine given intranasally once at least 30 minutes before anaesthetic induction
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 4 mcg/kg (Active Comparator): 4 mcg/kg dexmedetomidine given intranasally once at least 30 minutes before anaesthetic induction
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Either 2mcg/kg or 4mcg/kg of intranasal dexmedetomidine will be given to assess efficacy of preoperative sedation
  Other Names: Precedex

SUMMARY:
The purpose of the study is to determine if 4mcg/kg of intranasal dexmedetomidine is better than 2mcg/kg in successfully sedating a child prior to induction of anesthesia.

DETAILED DESCRIPTION:
Dexmedetomidine is a selective alpha-2 adrenoreceptor agonist that has sedative, anxiolytic and analgesic properties without causing respiratory depression. It has been administered safely and effectively via a number of routes including as an intravenous infusion, intramuscularly, intranasally, buccally and orally .

Yuen et al established that the median time of onset of sedation is 25-30 minutes, making it an ideal agent for preoperative sedation. The same group also studied doses of 1 mcg/kg and 2 mcg/kg as a sedative premedication and found that the success rates of appropriate sedation at induction in children aged 1 to 8 years were 53% and 66% respectively, with a dose related increase in successful sedation.

Much higher doses of dexmedetomidine have also been used safely. Administered intravenously, 3mcg/kg of dexmedetomidine has been shown to provide satisfactory sedation for paediatric MRI in 97% of cases, without adverse effects.

The investigators aim to show that high dose intranasal dexmedetomidine is a safe, effective and an easily administered sedative premedication.

The investigators hypothesise that 4mcg/kg compared to 2mcg/kg of intranasal dexmedetomidine will lead to at least a 20% increase in the proportion of satisfactorily sedated patients at the time of anaesthesia induction.

The primary outcome will be the proportion of children with satisfactory sedation at the time of anaesthesia induction.

Suitable patients will be identified from the theatre lists and consent will be sought from their legal guardians during preassessment clinic or during their anaesthetic preoperative assessment on the ward.

In a previous study, 66% of children aged 1-5 years were satisfactorily sedated at the time of induction with 2 mcg/kg of intranasal dexmedetomidine. In order to find a 20% difference with 4 mcg/kg of dexmedetomidine, the investigators' sample size needs to be 140 (70 in each group), for a power of 0.8 and a 5% false positive rate.

The demographic data will be analysed by t test and chi-square test. The proportions of satisfactory sedation will be analysed by chi-square test. The onset sedation time and duration of sedation will be analysed by survival analysis. The vital signs over times will be expressed by percentage changes from baseline and estimated by mean and standard errors. A p-value<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All children of American Society of Anesthesiologists (ASA) physical status classification I or II (healthy) between the ages of 6 months and 5 years undergoing surgery at Queen Mary Hospital

Exclusion Criteria:

* Any patient receiving other sedative premedication, allergy to dexmedetomidine, organ dysfunction, cardiac arrhythmia and congenital heart disease.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Satisfactory sedation | From 30 minutes post drug administration to induction of anaesthesia (average 30 minutes)
  The primary outcome will be the proportion of children with satisfactory sedation at the time of anaesthesic induction.

SECONDARY OUTCOMES:
Time to satisfactory sedation | From time of drug administration to when Observer's Assessment of Alertness/ Sedation Score is 2 or less (from 0 minutes to 30 minutes)
  Time taken from drug administration to when the child's sedation level is that of only responding after mild prodding or shaking
Blood pressure | From drug administration to end of anaesthesia (on average 1 to 3 hours)
  Blood pressure will be taken every 5 minutes
Heart rate | From drug administration to end of anaesthesia (on average 1 to 3 hours)
  Heart rate will be taken every 5 minutes
Oxygen saturations | From drug administration to end of anaesthesia (on average 1 to 3 hours)
  Oxygen saturations will be taken every 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sophie E Liu, MBBS, Principal Investigator — Hong Kong University
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Result] Pestieau SR, Quezado ZM, Johnson YJ, Anderson JL, Cheng YI, McCarter RJ, Choi S, Finkel JC. High-dose dexmedetomidine increases the opioid-free interval and decreases opioid requirement after tonsillectomy in children. Can J Anaesth. 2011 Jun;58(6):540-50. doi: 10.1007/s12630-011-9493-7. Epub 2011 Apr 2. PMID 21461792
- [Result] Mason KP, Zurakowski D, Zgleszewski SE, Robson CD, Carrier M, Hickey PR, Dinardo JA. High dose dexmedetomidine as the sole sedative for pediatric MRI. Paediatr Anaesth. 2008 May;18(5):403-11. doi: 10.1111/j.1460-9592.2008.02468.x. Epub 2008 Mar 18. PMID 18363626
- [Result] Mason KP, Lubisch NB, Robinson F, Roskos R. Intramuscular dexmedetomidine sedation for pediatric MRI and CT. AJR Am J Roentgenol. 2011 Sep;197(3):720-5. doi: 10.2214/AJR.10.6134. PMID 21862817
- [Result] Yuen VM, Irwin MG, Hui TW, Yuen MK, Lee LH. A double-blind, crossover assessment of the sedative and analgesic effects of intranasal dexmedetomidine. Anesth Analg. 2007 Aug;105(2):374-80. doi: 10.1213/01.ane.0000269488.06546.7c. PMID 17646493
- [Result] Yuen VM, Hui TW, Irwin MG, Yao TJ, Chan L, Wong GL, Shahnaz Hasan M, Shariffuddin II. A randomised comparison of two intranasal dexmedetomidine doses for premedication in children. Anaesthesia. 2012 Nov;67(11):1210-6. doi: 10.1111/j.1365-2044.2012.07309.x. Epub 2012 Sep 5. PMID 22950484